CLINICAL TRIAL: NCT04596358
Title: Interplay Between Adherence to the Mediterranean Diet, Lipid Profile and Blood Pressure: a Comparative Survey Among Healthcare and Non-Healthcare Female Workers
Status: Completed | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Collaborators: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Antonella Pipoli, Medical Doctor, University of Bari Aldo Moro
Other Study IDs: 10/2018
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diet Habit; Hypercholesterolemia; Hypertension
Keywords: Mediterranean Diet; Lipid profile; Healthcare workers
MeSH Terms: conditions — Feeding Behavior; Hypercholesterolemia; Hypertension | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healtcare workers: Women who work as nurses or doctors in public hospitals of which anthropometric and haematochemical data have been collected. Workers were given a questionnaire for the evaluation of the adherence to the Mediterranean diet.
  Interventions: Other: Observational
- Non-Healthcare workers: Women who perform technical and managerial professions in a public administration body of which anthropometric and haematochemical data have been collected. Workers were given a questionnaire for the evaluation of the adherence to the Mediterranean diet.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Evaluation of adherence to the Mediterranean diet through the administration of the Med Diet Score questionnaire.

SUMMARY:
The study aims at testing the level of adherence to the Mediterranean diet among health-workers, comparing this aspect to the extra-working physical activity, anthropometric measures and prevalence of cardiovascular, metabolic and neoplastic diseases previously diagnosed.

DETAILED DESCRIPTION:
The study had a cross-sectional setting and included employees of both genders currently in service.

Baseline data collection was structured as follows:

* Clinical assessment and pathological history
* Anthropometric measurements;
* Haematochemical examinations;
* Screening to adherence to Med-Diet by using "MedDietScore" questionnaire
* Assessment of the Harvard Cancer Risk Index for the evaluation of risk factors, modifiable and not, of the most frequent oncological diseases in Italy (colon, lung, breast and prostate). The index provides an estimate of individual cancer risk and is not equivalent to a cancer diagnosis. In addition, the Harvard Cancer Risk Index itself can allow the doctor to advise the worker on useful measures to reduce it;
* International Physical Activity Questionnairre (IPAQ)
* Major anthropometric and haematochemical data also allow to obtain one of the most used risk indexes for cardiovascular diseases in the scientific literature the Framingham Score.

ELIGIBILITY:
Inclusion Criteria:

* Women of working age
* Level of education at least equal to Bachelor's degree

Exclusion Criteria:

* Men
* Women under 20 years old or over 65 years old

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: One hundred and forty-seven subjects were randomly recruited at the Operating Unit of Occupational Medicine of the University Polyclinic Hospital of Bari in the last quarter of 2019. The whole sample included only female employees of public companies with at least 16 years of schooling, and subject to health surveillance by the occupational physicians of the above Operating Unit, subdivided as follows: fifty-nine HCWs (doctors and professional nurses) employees at the University Hospital of Bari, and eighty-eight employees of other public companies but not operating in the field of healthcare (non-HCWs).
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet greater control of circulating lipid levels | at Baseline
  Score of adherence (points)

SECONDARY OUTCOMES:
Fasting plasma glucose | Baseline
  Fasting plasma glucose in mg/dl
Serum insulin | Baseline
  Serum insulin microU/ml
systolic blood pressure | Baseline
  systolic blood pressure (mmHg)
diastolic blood pressure | Baseline
  diastolic blood pressure (mmHg)
Waist circumference | Baseline
  Waist circumference in centimeters
BMI (Body Mass Index) | Baseline
  BMI in kilograms/(meters)2
LDL-Cholesterol | Baseline
  LDL-Cholesterol in mg/dl
Triglycerides | Baseline
  Triglyceridesin mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Antonella Pipoli, Bari, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menotti A, Kromhout D, Blackburn H, Fidanza F, Buzina R, Nissinen A. Food intake patterns and 25-year mortality from coronary heart disease: cross-cultural correlations in the Seven Countries Study. The Seven Countries Study Research Group. Eur J Epidemiol. 1999 Jul;15(6):507-15. doi: 10.1023/a:1007529206050. PMID 10485342
- [Background] D'Alessandro A, De Pergola G. Mediterranean diet pyramid: a proposal for Italian people. Nutrients. 2014 Oct 16;6(10):4302-16. doi: 10.3390/nu6104302. PMID 25325250
- [Background] Di Lorenzo L, Pipoli A, Manghisi NM, Clodoveo ML, Corbo F, De Pergola G, Sabba C. Nutritional hazard analysis and critical control points at work (NACCPW): interdisciplinary assessment of subjective and metabolic work-related risk of the workers and their prevention. Int J Food Sci Nutr. 2020 Nov;71(7):902-908. doi: 10.1080/09637486.2020.1750572. Epub 2020 Apr 7. PMID 32255377
- [Background] Juarez-Perez CA, Aguilar-Madrid G, Haro-Garcia LC, Gopar-Nieto R, Cabello-Lopez A, Jimenez-Ramirez C, Aguado A, Martinez-Mendez LM, Chavez-Negrete A. Increased Cardiovascular Risk Using Atherogenic Index Measurement Among Healthcare Workers. Arch Med Res. 2015 Apr;46(3):233-9. doi: 10.1016/j.arcmed.2015.03.002. Epub 2015 Mar 19. PMID 25797688
- [Background] Panagiotakos DB, Pitsavos C, Stefanadis C. Dietary patterns: a Mediterranean diet score and its relation to clinical and biological markers of cardiovascular disease risk. Nutr Metab Cardiovasc Dis. 2006 Dec;16(8):559-68. doi: 10.1016/j.numecd.2005.08.006. Epub 2006 Feb 9. PMID 17126772
- [Derived] Di Lorenzo L, Vimercati L, Pipoli A, Manghisi NM, Lampignano L, Caputi A, De Maria L, Zupo R, De Pergola G. Interplay Between Adherence to the Mediterranean Diet and Lipid Profile: A Comparative Survey Between Day-Time Healthcare and Non-healthcare Female Workers. Front Public Health. 2021 Nov 4;9:649760. doi: 10.3389/fpubh.2021.649760. eCollection 2021. PMID 34805058